CLINICAL TRIAL: NCT00269022
Title: A Single Blind, Placebo Controlled, Multi-Centre Study to Investigate the Pharmacokinetics, Safety, Tolerability and Pharmacodynamics of the TRPV1 Antagonist SB-705498 Against the Pain of Acute Migraine.
Brief Title: Use Of SB-705498 In The Acute Treatment Of Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SB-705498/008
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Migraine, Acute
Keywords: SB-705498 acute migraine single dose TRPV1 combination inpatient outpatient study
MeSH Terms: conditions — Migraine Disorders | interventions — SB 705498

INTERVENTIONS:
Drug: SB-705498

SUMMARY:
Despite the success of the triptan class of drugs, approximately 60% of patients who take medication at the moderate to severe pain stage of acute migraine, still have pain of mild or greater degree at 2 hrs post dose. SB-705498 is a novel, first in class TRPV1 receptor antagonist under development for the treatment of migraine pain. Preclinical experiments have demonstrated that the TRPV1 receptor is expressed both centrally and peripherally in the trigeminal system and inhibition of TRPV1 with SB-705498 can both prevent and reverse established central sensitisation.

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects suffering from moderate to severe migraine headache with or without aura.
* Women of child bearing potential must use an effective method of contraception.
* Have had at least a 1 year history of migraine and the age of onset was prior to 50 years.
* Suffering 1 to 6 migraine attacks per month for at least the last 3 months and should have at least 48 hours free of headache between migraine attacks.

Exclusion criteria:

* Headache for 15 days/month or greater in any of the three months (90 days) preceding entry into the study.
* Use of migraine medications (e.g., ergotamine, triptan, opioid, or combination medication) on >/= 10 days per month on a regular basis for >/= 3 months.
* Use of analgesics >/=15 days per month for >/=3 months, uses an opiate (except codeine) as first line treatment for migraine.
* Migraine symptoms do not respond to any of the triptan drugs (e.g., Imitrex, Relpax, Maxalt).
* Have uncontrolled hypertension or a history/ presence of multiple cardiovascular risk factors such as, but not limited to family history, myocardial infarction, coronary artery disease, vasospastic angina, heart failure, cardiac arrhythmias or history or presence of cerebrovascular disease, including transient ischemic attack, stroke or peripheral arterial disease.
* History of alcohol, substance or drug abuse within the last year.
* Participation in a trial with a new chemical entity within 3 months before the start of the study.
* Participation in any other research trial within 30 days prior to the first dose of current study medication is not permitted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2006-01

PRIMARY OUTCOMES:
Percentage of subjects who are pain free at 2 hrs post-dose (e.g., have moderate to severe pain at baseline and no pain at 2 hrs post-dose).

SECONDARY OUTCOMES:
Pain free at 30mins, 1,3,4,5&6hrs Headache relief and absence/presence of associated symptoms at 30 mins, 1,2,3,4,5&6hrs Additional migraine medication Safety tests ( e.g., continuous ECG, laboratory tests) Heat pain thresholds.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Randwick, New South Wales, Australia
- GSK Investigational Site, Toronto, Ontario, Canada
- GSK Investigational Site, Leiden, Netherlands
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom